CLINICAL TRIAL: NCT01790880
Title: Enhancing Written Communication in Persons With Aphasia: A Clinical Trial
Brief Title: Enhancing Written Communication in Persons With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Leora Cherney, Senior Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 74374
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Stroke; Speech Rehabilitation
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORLA (Active Comparator): Practice on ORLA (Oral Reading for Language in Aphasia), a computer-based virtual therapy system, for 90 minutes per day, 6 days per week for 6 weeks.
  Interventions: Behavioral: ORLA
- ORLA + Writing (Experimental): Practice on "ORLA + writing" computer program, 90 minutes per day, 6 days per week, for 6 weeks.
  Interventions: Behavioral: ORLA + Writing

INTERVENTIONS:
Behavioral: ORLA — Practice on ORLA (Oral Reading for Language in Aphasia), a computer-based virtual therapy system.
  Arms: ORLA
Behavioral: ORLA + Writing — Treatment includes writing of sentences in combination with ORLA
  Arms: ORLA + Writing

SUMMARY:
The purpose of this study is to evaluate whether a computerized speech-language treatment delivered by a virtual therapist (Oral Reading for Language in Aphasia (ORLA) + Writing) results in improved written communication skills of study participants with aphasia (i.e., difficulty with the comprehension and expression of spoken and written language).

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the most common cause of disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. Approximately 150,000 to 250,000 stroke survivors becoming severely and permanently disabled each year. A common neurological deficit among stroke survivors, and thus a substantial contributor to post-stroke disability, is aphasia. The loss of, or difficulty with language is extremely debilitating.

Adequate written communication skills may be one of the barriers that has prevented individuals with aphasia from returning to work. Writing skills are also important for participation in social roles, such as household management, civic activities, or recreational activities with friends. Individuals with aphasia struggle to compose written documents such as personal letters, memos and reports. Furthermore, society's increased reliance on written forms of communication including email correspondence, instant messaging, texting, Twitter, and social networking sites such as Facebook, exacerbate the challenge that individuals with aphasia have in connecting with others, reestablishing and redefining their social roles and accomplishing their life-participation goals.

Computer-directed treatment offers a practical alternative to one-on-one traditional treatment provided by a clinician and may be a cost-effective way of extending therapy beyond the hospital and clinic to meet the needs of the growing numbers of individuals with chronic aphasia and to help them reintegrate into the community and workforce. This project evaluates the efficacy of a theoretically-motivated writing program that has been integrated with novel computer-based virtual therapy systems and that can be provided intensively to individuals with chronic aphasia.

ELIGIBILITY:
Inclusion Criteria:

1. men or women with diagnosis of an aphasia subsequent to a left-hemisphere infarct(s) that is confirmed by CT scan or MRI
2. an Aphasia Quotient score on the Western Aphasia Battery of 50-85.
3. 6 months post injury
4. premorbidly right handed, determined by Edinburgh Handedness Inventory
5. completed at least an eighth grade education
6. premorbidly literate in English
7. visual acuity may be corrected but must be sufficient for reading visual stimuli on computer screen
8. auditory acuity may be aided but must be sufficient for hearing auditory stimuli in ORLA program

Exclusion Criteria:

1. any other neurological condition (other than cerebral vascular disease) that could potentially affect cognition or speech, such as Parkinson's Disease, Alzheimer's Dementia, traumatic brain injury.
2. any significant psychiatric history prior to the stroke, such as severe major depression or psychotic disorder requiring hospitalization; subjects with mood disorders who are currently stable on treatment will be considered.
3. active substance abuse.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2017-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Writing Score on the Western Aphasia Battery-Revised (WAB-R) from pre-treatment to post-treatment | Change from baseline to 6 weeks

SECONDARY OUTCOMES:
Western Aphasia Battery-Revised Aphasia Quotient (WAB-R AQ) | Change from baseline to 6 weeks
Written Language Sample Analysis | Change from baseline to 6 weeks
  Written responses on the Picture Description task of the Western Aphasia Battery-Revised and on a written picture-sequenced story retelling task will be scored for Correct Information Units
Communicative Effectiveness Index (CETI) | Change from baseline to 6 weeks
ASHA Quality of Communication Life Scale (QCL) | Change from baseline to 6 weeks
Community Integration Questionnaire (CIQ) | Change from baseline to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Aphasia Research and Treatment, Rehabilitation Institute of Chicago, Chicago, Illinois, United States